CLINICAL TRIAL: NCT00463970
Title: A Randomized Controlled Multicentre Trial of a Brief Intervention (BI) Versus a BI Plus Cognitive Behavioural Treatment (CBT) Versus Nutritional Supplementation for Patients With Long-lasting Back Pain.
Brief Title: Cognitive Interventions and Nutritional Supplementation for Patients With Long-lasting Back Pain
Acronym: CINS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: The Research Council of Norway (Other); University of Bergen (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CINS2007
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Brief cognitive intervention; Cognitive behavior therapy; Seal oil
MeSH Terms: interventions — Crisis Intervention; Cognitive Behavioral Therapy; Cognitive Training; Geologic Sediments; Dietary Supplements; Soybean Oil; Plant Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Brief Intervention
  Interventions: Behavioral: Brief Intervention
- 2 (Experimental): Cognitive Behavioural Therapy
  Interventions: Behavioral: Cognitive Behavioural Therapy
- 3 (Experimental): Seal oil
  Interventions: Dietary Supplement: Seal oil
- 4 (Placebo Comparator): Soy oil
  Interventions: Dietary Supplement: Soy oil

INTERVENTIONS:
Behavioral: Brief Intervention — Physical examination, education and follow up by a physiotherapist
  Other Names: Brief Education; Light mobilization treatment
  Arms: 1
Behavioral: Cognitive Behavioural Therapy — 7 sessions of CBT over a period of 2 months, included a booster session after 3 months
  Other Names: Cognitive behavioral treatment; Cognitive rehabilitation
  Arms: 2
Dietary Supplement: Seal oil — 20 capsules per day for 3 months
  Other Names: Marine oil; Nutritional supplement
  Arms: 3
Dietary Supplement: Soy oil — 20 capsules per day for 3 months
  Other Names: Vegetable oil; Nutritional supplement
  Arms: 4

SUMMARY:
CINS is a large multicentre study which aims to test out the effect of 4 different interventions, namely a brief cognitive intervention (BI), a more extensive cognitive behavioural intervention (CBT), and 2 different nutritional supplementations (seal oil and soy oil) in a population of chronic low back pain patients sicklisted for 2-10 months.

DETAILED DESCRIPTION:
The treatment principles for low back pain, and also other types of non-specific muscle pain, have changed dramatically over the last 10 to 15 years; from traditional treatment like bed rest and inactivity to more active treatment strategies ("the back pain revolution"; Waddell et al 1997). Norwegian research has been in the forefront, particularly in demonstrating the clinical and cost effective brief interventions (BI) (Indahl et al., 1995, 1998; Hagen et al 2000, 2004, Brox et al 2003, Storheim et al 2003). However, about 30% of the patients do not recover or return to normal social and working life. The aim of this study is therefore to see if a longer cognitive behavioural intervention (CBT) has an additional benefit to BI, and to compare this with a potentially beneficial dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* Patients sicklisted 2-10 months for low back pain
* The following diagnosis are included: L02, L03, L84 and L86

Exclusion Criteria:

* Being off the sick list
* Pregnancy
* Osteoporosis
* Cancer
* L diagnoses suggesting recent low back pain trauma
* Specific spinal or other injuries which may account for the current back pain
* Serious psychiatric pathology

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 414 (Actual)
Dates: Start 2008-02; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sickness leave | 2008-2020

SECONDARY OUTCOMES:
Health complaints | 2008-2010
Psychopathology | 2008-2010
Cortisol curves | 2008-2010
Function | 2008-2010

CONTACTS AND LOCATIONS:
Overall Officials: Hege R Eriksen, Professor, Principal Investigator — Unifob health, University of Bergen
Locations (2):
- Norway (2):
  - Uni Research Health, Bergen
  - Torill H Tveito, Bergen

REFERENCES:
- [Result] Reme SE, Tveito TH, Chalder T, Bjorkkjaer T, Indahl A, Brox JI, Fors E, Hagen EM, Eriksen HR. Protocol for the Cognitive Interventions and Nutritional Supplements (CINS) trial: a randomized controlled multicenter trial of a brief intervention (BI) versus a BI plus cognitive behavioral treatment (CBT) versus nutritional supplements for patients with long-lasting muscle and back pain. BMC Musculoskelet Disord. 2011 Jul 7;12:152. doi: 10.1186/1471-2474-12-152. PMID 21736730
- [Result] Reme SE, Tangen T, Moe T, Eriksen HR. Prevalence of psychiatric disorders in sick listed chronic low back pain patients. Eur J Pain. 2011 Nov;15(10):1075-80. doi: 10.1016/j.ejpain.2011.04.012. Epub 2011 May 17. PMID 21592832
- [Result] Harris A, Endresen Reme S, Tangen T, Hansen AM, Helene Garde A, Eriksen HR. Diurnal cortisol rhythm: Associated with anxiety and depression, or just an indication of lack of energy? Psychiatry Res. 2015 Aug 15;228(2):209-15. doi: 10.1016/j.psychres.2015.04.006. Epub 2015 Apr 24. PMID 26001959
- [Result] Reme SE, Tveito TH, Harris A, Lie SA, Grasdal A, Indahl A, Brox JI, Tangen T, Hagen EM, Gismervik S, Odegard A, Fr Yland L, Fors EA, Chalder T, Eriksen HR. Cognitive Interventions and Nutritional Supplements (The CINS Trial): A Randomized Controlled, Multicenter Trial Comparing a Brief Intervention With Additional Cognitive Behavioral Therapy, Seal Oil, and Soy Oil for Sick-Listed Low Back Pain Patients. Spine (Phila Pa 1976). 2016 Oct 15;41(20):1557-1564. doi: 10.1097/BRS.0000000000001596. PMID 27760062
- [Derived] Opsahl J, Eriksen HR, Tveito TH. Do expectancies of return to work and Job satisfaction predict actual return to work in workers with long lasting LBP? BMC Musculoskelet Disord. 2016 Nov 17;17(1):481. doi: 10.1186/s12891-016-1314-2. PMID 27855684
- See also: Study website — http://uni.no/nb/uni-helse/stress-helse-og-rehabilitering/ryggstudien-cins/